CLINICAL TRIAL: NCT04922359
Title: Effect of Perioperative Lidocaine on Gastrointestinal Function Recovery After Lumbar Spine Surgery in Adults: a Multicenter, Randomized, Double-blind, Controlled Study
Brief Title: Effect of Perioperative Lidocaine on Gastrointestinal Function Recovery After Lumbar Spine Surgery in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Wangjing Hospital, China Academy of Chinese Medical Sciences (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Head of Anesthesiology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021PHB059-001
Record Dates: First submitted 2021-06-06; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Spinal Surgery; Lidocaine; Pain; Opioid Consumption; Gastrointestinal Dysfunction
Keywords: Lidocaine; Gastrointestinal Dysfunction; Spinal surgery; Opioid consumption
MeSH Terms: conditions — Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Lidocaine group (Experimental)
  Interventions: Drug: Lidocain
- Placebo Comparator: comparator group (Placebo Comparator)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Lidocain — Patients received 1.5mg/kg of intravenous lidocaine during induction of anesthesia and 1.5 mg/kg/h for anesthesia maintenance.
  Arms: Experimental: Lidocaine group
Drug: normal saline — Patients received 0.075ml/kg of intravenous normal saline during induction of anesthesia and 0.075ml/kg/h for anesthesia maintenance.
  Arms: Placebo Comparator: comparator group

SUMMARY:
Spinal surgery often involves multiple segments. The trauma of surgery is large, the duration of postoperative pain is long, and the pain is severe. Therefore, the use of opioids in perioperative period is large. Although the application of * large amounts of opioids can effectively inhibit pain, it will delay the recovery of urine retention, sedation, respiratory depression and gastrointestinal function. The delayed recovery of gastrointestinal function will increase the postoperative complications, and then increase the length of hospital stay and the cost of patients. Therefore, reducing the dosage of opioids to promote the recovery of gastrointestinal function has become the research direction. Intravenous lidocaine has been proved to be effective in reducing the dosage of opioids during the perioperative period of gastrointestinal surgery and promoting the recovery of postoperative gastrointestinal function. However, there are few studies on the application of lidocaine during the perioperative period of spinal surgery, especially the impact on postoperative gastrointestinal function. In this study, a multicenter, randomized, double-blind, controlled study was conducted to explore the effect of perioperative lidocaine on the recovery of gastrointestinal function after adult lumbar surgery. We hypothesized that lidocaine could shorten the recovery time of gastrointestinal function after lumbar surgery

ELIGIBILITY:
Inclusion Criteria:

1. age 60 to 80;
2. ASA physical status score of I, II or III;
3. Scheduled to undergo a posterior lumbar surgery;
4. Ideal body weight≤80 kg;

Exclusion Criteria:

1. Those who are refused to be included;
2. Those who are allergic to the drugs used in this study;
3. Emergency operation
4. Degree II or III atrioventricular block
5. heart failure
6. History of ALS, preexcitation or active dysrhythmia
7. Severe liver injury (bilirubin > 1.46 mg/dl)
8. Severe renal injury (creatinine clearance < 30 ml/min) or Renal failure
9. History of epilepsy
10. History of porphyria
11. Preoperative hypotension (SBP< 90mmHg)
12. Drug contraindications of NSAIDs
13. Allergic to anaesthetic

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
First anal exhaust time | Day 0
  Time of first anal exhaust after operation

SECONDARY OUTCOMES:
First defecation time | Day 0
  Time of first defecation after operation
First diet time | Day 0
  Time of first feeding after operation
Time to get out of bed | Day 0
  Time to get out of bed after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China